CLINICAL TRIAL: NCT06208033
Title: A Single-arm, Sequential Study Assessing the Efficacy and Safety of SMET12 and Toripalimab Combined Chemotherapy in Patients With EGFR Positive Advanced Non-small Cell Lung Cancer (NSCLC) : First-line Treatment or Failed From First-line Immune Checkpoint Inhibitor Treatment.
Brief Title: SMET12 and Toripalimab Combined Chemotherapy in Patients With EGFR Positive Advanced Non-small Cell Lung Cancer (NSCLC)
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCOG009
Record Dates: First submitted 2024-01-05; First posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: EGFR Positive Non-small Cell Lung Cancer
MeSH Terms: interventions — toripalimab; Pemetrexed; Carboplatin; Paclitaxel; Cisplatin; Docetaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment-naïve subjects with EGFR positive advanced Lung Adenocarcinoma (Experimental): toripalimab：3mg/kg， Q2W； SMET12：60μg，Q2W； Pemetrexed Disodium 500mg/m2 d+Carboplatin AUV＝5 d1 Q3W，administered for 2~4 cycles
  Interventions: Drug: SMET12
- Treatment-naïve subjects with EGFR positive advanced Lung Squamous Cell Carcinoma (Experimental): toripalimab：3mg/kg， Q2W； SMET12：60μg，Q2W； paclitaxel 100mg/m2 d1，d8，d15+cisplatin 75mg/m2 d1 Q3W， administered for 2~4 cycles
  Interventions: Drug: SMET12
- Subjects resistant to first-line treatment contain immune checkpoint inhibitors (Experimental): toripalimab：3mg/kg， Q2W； SMET12：60μg，Q2W； Docetaxel 60-75 mg/m2 d1Q3W，administered for 2~4 cycles
  Interventions: Drug: SMET12

INTERVENTIONS:
Drug: SMET12 — 1. platinum-containing two-drug chemotherapy：Carboplatin plus Pemetrexed Disodium, administrated for 2-4 cycles, three weeks for one cycyles;Carboplatin 500mg/m2 d1,Pemetrexed Disodium AUV＝5 d1,Q3W;
  2. Toripalimab, IV, 3mg/kg，Q2W；
  3. SMET12: IV，60μg，Q2W，injected the day after toripalimab ；
  Other Names: toripalimab; Pemetrexed Disodium; Carboplatin
  Arms: Treatment-naïve subjects with EGFR positive advanced Lung Adenocarcinoma
Drug: SMET12 — 1. platinum-containing two-drug chemotherapy：Carboplatin plus Pemetrexed Disodium, administrated for 2-4 cycles, 3 weeks for one cycle.cisplatin 75mg/m2 d1 Q3W,paclitaxel 100mg/m2 d1，d8，d15;
  2. Toripalimab, IV, 3mg/kg，Q2W；
  3. SMET12: IV，60μg，Q2W，injected the day after toripalimab ；
  Other Names: toripalimab; paclitaxel; cisplatin
  Arms: Treatment-naïve subjects with EGFR positive advanced Lung Squamous Cell Carcinoma
Drug: SMET12 — 1. chemotherapy：Docetaxel 60-75 mg/m2 d1, administrated for 2-4 cycles, 3 weeks for one cycle.
  2. Toripalimab, IV, 3mg/kg，Q2W；
  3. SMET12: IV，60μg，Q2W，injected the day after toripalimab ；
  Other Names: toripalimab; Docetaxel
  Arms: Subjects resistant to first-line treatment contain immune checkpoint inhibitors

SUMMARY:
This is a single-arm, sequential study assessing the efficacy and safety of SMET12 and Toripalimab combined chemotherapy in patients with EGFR positive advanced non-small cell lung cancer (NSCLC) : first-line treatment or failed from first-line immune checkpoint inhibitor treatment.The primary objective is to evaluate the anti-tumor activity and safety of SMET12 and Toripalimab combined chemotherapy in patients with EGFR positive advanced NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* 1. Has fully understood and voluntarily signed an informed consent form for this study , willing and able to comply with study procedures.

  2. Age ≥ 18 years. 3. Histologically confirmed EGFR positive (immunohistochemistry ≥ [+]) advanced NSCLC ,including: (1) Cohort A: Treatment-naïve subjects; (2) Cohort B: Subjects resistant to first-line treatment contain immune checkpoint inhibitors (stability period > 3 months).

  4. At least one measurable lesion via RECIST v1.1 criteria 5. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1. 6. Expected survival ≥ 3 months. 7. Adequate organ function .

Exclusion Criteria:

* 1. Driver gene-positive (EGFR, ALK, ROS1) . 2. history of dual primary malignancies within the past 5 years. 3. active autoimmune diseases or a history of autoimmune disorders requiring systemic corticosteroid therapy.

  4. systemic infections requiring systemic treatment. 5. known central nervous system metastases or other central nervous system diseases or abnormalities deemed unsuitable for inclusion in this study by the investigator.

  6. Fertile individuals unable to maintain effective contraception during the trial.

  7. Subjects in Cohort B who have received prior docetaxel treatment. 8. Subjects in Cohort B who experienced Grade 3 or higher immune-related adverse events during first-line treatment with immune checkpoint inhibitors.

  9. Individuals deemed unsuitable for participation in this clinical trial by the investigator for various reasons .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-01-10 (Estimated); Primary Completion 2024-10-20 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
incidence of adverse events | 1 year
  Adverse events incidence refers to the frequency of adverse events
rate of adverse events | 1 year
  All adverse events will also be rated based on the NCI CTCAE version 5.0.
Laboratory aberrations | 1 year
  Laboratory outliers refer to measurement results that significantly deviate from the normal reference range in laboratory testing.

SECONDARY OUTCOMES:
disease control rate | 1 year
  Disease control rate: DCR
Progression-free survival | 1 year
  Progression-free survival (PFS) as assessed by the investigators according to RECIST 1.1 criteria
DOR（ Duration of Response） | 1 year
  Duration of response (DoR) is defined as the time from first confirmed response (complete response or partial response) to the date of the initial objectively documented tumor progression as determined per investigator assessment using RECIST 1.1 criteria or death due to any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Cancer Hospital, Fuzhou, China

REFERENCES:
- [Derived] Lin J, Chen S, Li M, Weng L, Xu H, Wang Q, Zhang J, Lin D, Wang H, Liu Q, He Z. Efficacy and safety of SMET12 in combination with toripalimab and chemotherapy in advanced non-small-cell lung cancer patients tested positive for EGFR protein who are treatment-naive or harbor acquired resistance to standard therapy: a phase 2, multi-cohort clinical trial. Front Immunol. 2026 Jan 8;16:1706961. doi: 10.3389/fimmu.2025.1706961. eCollection 2025. PMID 41583476